CLINICAL TRIAL: NCT05130333
Title: The Clinical Research of Needle Electrodes Used in Bispectral Index to Monitor the Depth of Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0582
Record Dates: First submitted 2021-11-03; First posted 2021-11-23 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-10

CONDITIONS: Intraoperative Monitoring; Depth of Anesthesia
Keywords: sedation; Needle electrodes; BIS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-cardiac surgery patients under general anesthesia: > 18y/o patients undergoing noncardiac surgery with BIS monitoring under general anesthesia.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In this study, the EEG information of patients was collected by different BIS electrodes, in order to compare the quality of EEG signals obtained by subdermal needle electrodes and the original BIS sensors, and try to use primitive EEG signals to develop a new calculation of needle electrode to monitor the depth of anesthesia.

DETAILED DESCRIPTION:
After the patient enters the room, non-invasive BP, HR, end-tidal CO2, SPO2 and other routine monitoring are performed, and the corresponding BIS electrodes are worn to the patient. The anesthesiologist decides whether to perform invasive hemodynamic monitoring, such as invasive arterial blood pressure monitoring, central venous pressure monitoring, etc., depending on the patient's condition and surgical requirements. The induction and maintenance of anesthesia is the routine scheme in the Second Affiliated Hospital of Zhejiang University , and the medication and dose are based on the judgment of the main anesthesiologist . After induction, endotracheal intubation was performed and mechanical ventilation was given. After anesthesia induction, install subcutaneous needle electrode to the patient. BIS values were collected using two BIS monitoring systems, one using the original BIS sensor and the other connected to the needle electrodes.During the operation, the anesthesiologist adjusted the depth of anesthesia according to the original BIS value, and propofol was used to improve the depth of sedation if the BIS value was greater than 60. In this study, surface acoustic wave electronic nose was used to monitor the exhaled propofol concentration of patients undergoing general anesthesia.The BIS value, hemodynamic information, exhaled propofol concentration and plasma propofol concentration were recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASAⅠ~Ⅲ
* Over 18 years old
* Patients undergoing General Anesthesia surgery requiring BIS Monitoring
* Obtained informed consent

Exclusion Criteria:

* Patients who have mental disorders and unable to answer
* Patients who have taken anti-epileptic drugs and psychotropic drugs for a long time
* Patients who are pregnant
* Patients who refuse to participate in this trial
* Patients considered by the investigator to be unsuitable for inclusion in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General anesthesia patients undergoing non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-11-29 (Estimated); Primary Completion 2022-10-22 (Estimated); Study Completion 2023-02-22 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient | Through study completion, an average of 2 year
  The correlation coefficient between the BIS value measured by the subdermal needle electrodes and the BIS value measured by the original BIS sensors

SECONDARY OUTCOMES:
Correlation between BIS values and OAA/S score | Through study completion, an average of 2 year
  Comparison of the correlation between BIS values measured by two kinds of electrodes and OAA/S
Correlation between BIS values and propofol concentration | Through study completion, an average of 2 year
  Correlation between BIS values measured by two kinds of electrodes and propofol concentration in blood From Exhaled Gas
Correlation between BIS values and blood pressure and heart rate | Through study completion, an average of 2 year
  Correlation between BIS values measured by two kinds of electrodes and blood pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided